CLINICAL TRIAL: NCT00962975
Title: A Study of Pegasys Monotherapy in Patients With Chronic Hepatitis B Who Have Participated in Previous Studies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PP22612
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — dosage at discretion of investigator based on standard of care (180mcg sc weekly) for up to 48 weeks

SUMMARY:
In this open-label multicenter study the long-term effect of Pegasys monotherapy on pharmacodynamic HBV-related markers will be investigated in patients with chronic hepatitis B. Eligible patients will have completed treatment on another donor protocol (e.g. PP22512) and will receive Pegasys at an appropriate dose based on the standard of care (180mcg sc once weekly) for up to 48 weeks. Target sample size is <100.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >/=18 years of age
* previous participation in other donor protocol
* chronic hepatitis B
* no other anti-HBV treatment after completion of previous donor protocol
* female patients and female partners of male patients must use at least two methods of contraception until 28 days after completion of study

Exclusion Criteria:

* hepatic decompensation (Child-Pugh class B and C)
* antiviral, antineoplastic or immunomodulatory treatment
* evidence of alcohol and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The longitudinal effect on HBV-related markers: viral load, viral antigen/antibody, viral sequence, cellular and humoral immune responses, RNA | assessed every 2 months on treatment (not exceeding maximum approved duration), and up to week 24 of follow-up

SECONDARY OUTCOMES:
Safety and tolerability: AEs, laboratory parameters, vital signs, concomitant medications | assessed every 2 months on treatment and up to week 24 of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (2):
  - Los Angeles, California
  - San Francisco, California
- Grafton, New Zealand
- Singapore, Singapore
- Taipei, Taiwan